CLINICAL TRIAL: NCT00724711
Title: A Prospective, Randomized, Open Label Phase IV Study to Evaluate the Rationale of Switching From Fixed Dose Abacavir (ABC)/Lamivudine (3TC) to Fixed Dose Tenofovir DF (TDF)/Emtricitabine (FTC) in Virologically Suppressed, HIV-1 Infected Patients Maintained on a Ritonavir Boosted Protease Inhibitor Containing Antiretroviral Regimen
Brief Title: Safety and Efficacy Study of Switching From Epzicom to Truvada
Acronym: SWIFT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-164-0216
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infection
Keywords: HIV; HIV 1
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir; abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FTC/TDF (Truvada [TVD]) + PI/r (Experimental): Participants in this group received fixed-dose combination FTC 200 mg/TDF 300 mg (Truvada [TVD]) for 48 weeks. The prestudy ritonavir-boosted PI was continued unmodified through the 48 weeks of the study.
  Interventions: Drug: emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF)
- ABC/3TC + PI/r (Active Comparator): Participants in this group continued their prestudy therapy - ABC 600 mg/3TC 300 mg administered as one tablet orally once daily (Epzicom) plus ritonavir-boosted PI regimen, given orally for 48 weeks.
  Interventions: Drug: abacavir (ABC)/lamivudine (3TC)

INTERVENTIONS:
Drug: emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) — FTC 200 mg/TDF 300 mg tablet, once a day
  Other Names: Truvada
  Arms: FTC/TDF (Truvada [TVD]) + PI/r
Drug: abacavir (ABC)/lamivudine (3TC) — ABC 600 mg/3TC 300 mg tablet, once a day
  Other Names: Epzicom, Kivexa
  Arms: ABC/3TC + PI/r

SUMMARY:
This protocol describes a prospective, randomized, open-label, multicenter study to evaluate the safety and efficacy of switching from fixed dose abacavir (ABC)/lamivudine (3TC) to fixed dose emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) in virologically suppressed, human immunodeficiency virus type 1 (HIV-1) infected subjects maintained on a ritonavir-boosted protease inhibitor (PI/r)-containing antiretroviral (ARV) regimen. Duration of treatment is 48 weeks.

DETAILED DESCRIPTION:
This protocol describes a prospective, randomized, open-label, multicenter study to evaluate the safety and efficacy of switching from fixed dose ABC/3TC to fixed dose FTC/TDF in virologically suppressed, HIV-1 infected subjects maintained on a PI/r-containing ARV regimen.

Subjects were stratified based on the PI/r (ie, lopinavir/ritonavir [LPV/r] versus other boosted PIs) in their regimen, and the presence versus absence of comorbidities at screening (diabetes mellitus or cardiovascular disease such as hypertension, coronary artery disease, hyperlipidemia, history of myocardial infarction, cardiomyopathy, valvular heart disease, congenital heart disease, stroke, peripheral vascular disease, or arrhythmias). Subjects were randomized 1:1 to switch to FTC/TDF+PI/r or to continue on their existing regimen.

Subjects received study treatment for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult (greater than or equal to 18 years) males or non-pregnant, non-lactating females
* HIV-1 infected subjects currently receiving a ritonavir-boosted protease inhibitor and fixed-dose ABC/3TC regimen continuously for greater than or equal to 3 months
* HIV infection as documented by a validated HIV antibody enzyme-linked immunosorbent assay (ELISA) and confirmed by one of the following:

  * Immunoblot detection of HIV antibody
  * Positive HIV-1 blood culture
  * Positive HIV-1 serum P24 antigen
  * HIV-1 plasma viremia greater than 1000 copies/mL by polymerase chain reaction (PCR) or branched-chain deoxyribonucleic acid (bDNA) method
  * Detection of proviral DNA by PCR

(If confirmation of HIV infection is not available then repeat testing of HIV antibody will be required)

* Two consecutive plasma HIV-1 RNA concentration less than 200 copies/mL. The two HIV-1 RNA determinations ensure that the subject has been virologically-suppressed for at least 3 months prior to study entry:

  * The subject must have a plasma HIV-1 RNA level less than 200 copies/mL using the AmpliPrep/Taqman HIV-1 Test or Roche Amplicor HIV-1 Monitor Test Version 1.5 Ultrasensitive method at least 3 months prior to the screening visit, as the "qualifying HIV-1 RNA."
  * HIV-1 RNA less than 200 copies/mL measured by bDNA (Chiron 3.0) may be used as a qualifying HIV-1 RNA for entry to the study but not for the confirmatory HIV-1 RNA.
  * The subject must have a confirmed second plasma HIV-1 RNA less than 200 copies/mL at screening, as the "confirmatory HIV-1 RNA."
  * The subject must not have a plasma HIV-1 RNA greater than or equal to 200 copies/mL between the qualifying and confirmatory HIV-1 RNA measurements.
* Subjects receiving lipid-lowering agents (LLA) will be allowed; however, LLAs must be stable for greater than or equal to 3 months prior to study entry.
* Adequate renal function defined as a calculated CLcr greater than or equal to 50 mL/min according to the Cockcroft-Gault formula
* Negative serum pregnancy test (females of childbearing potential only)
* Hepatic transaminases alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 5 X upper limit of normal
* Males and females (of childbearing potential, ie, a non-menopausal female or a female with menopause < 2 years, and who has not had a hysterectomy, bilateral oophorectomy, or medically documented ovarian failure; this definition includes a young woman who has not yet started menstruating), and must agree to avoid pregnancy by sexual abstinence, or utilization of a highly effective method of birth control throughout the study period and for 30 days following discontinuation of study drug
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures

Exclusion Criteria:

* Subjects receiving ABC/3TC and a PI without ritonavir
* Subjects receiving other ARV agents (eg, 2 protease inhibitors boosted with low-dose ritonavir (ie, "double-boosted PI regimens"), nonnucleoside reverse transcriptase inhibitors [NNRTIs], integrase inhibitors, TDF, or other nucleoside reverse transcriptase inhibitor [NRTIs]) in addition to ABC/3TC and a ritonavir-boosted protease inhibitor
* Have known resistance to any of the study agents at any time in the past including NRTI resistance mutations (including but not limited to K65R, L74V/I, M184V/I, or thymidine analog mutations) and/or PI resistance mutations
* A new acquired immunodeficiency syndrome (AIDS) defining condition diagnosed (with the exception of CD4 criteria) within 30 days of baseline
* Previous therapy with agents with systemic myelosuppressive, pancreatoxic, hepatotoxic or cytotoxic potential within 3 months of study start or the expected need for such therapy at the time of enrollment
* Proven or suspected acute hepatitis in the 30 days prior to study entry
* Anticipated need to initiate drugs during the study that are contraindicated with protease inhibitors (except upon approval by Gilead)
* Receiving ongoing therapy with any of the following (administration of any of the following medications must be discontinued at least 30 days prior to the Baseline visit and for the duration of the study period):

  * Nephrotoxic agents (aminoglycoside antibiotics, amphotericin B, cidofovir, cisplatin, foscarnet, intravenous pentamidine, other agents with significant nephrotoxic potential)
  * Adefovir dipivoxil
  * Probenecid
  * Systemic chemotherapeutic agents (ie, cancer treatment medications)
  * Systemic corticosteroids
  * Interleukin-2 (IL-2)
  * Investigational agents (except upon approval by Gilead)
* Pregnant or lactating subjects
* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication
* Current alcohol or substance abuse judged by the investigator to potentially interfere with subject adherence
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Subjects with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of baseline and are not anticipated to require systemic therapy during the study.
* Active, serious infections (other than HIV-1 infection) requiring parenteral antimicrobial therapy within 15 days prior to screening
* Prior history of significant renal or bone disease
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements
* Known hypersensitivity to the study drugs, the metabolites or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Fralich, MD, Study Director — Gilead Sciences
Locations (80):
- United States (73):
  - Health For Life Clinic, PLLC, Little Rock, Arkansas
  - Vista Medical Partners, Beverly Hills, California
  - AHF, Beverly Hills, California
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Center for Special Immunology, Fountain Valley, California
  - Living Hope Clinical Foundation, Long Beach, California
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Anthony M Mills, MD, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Tarzana Treatment Center, Northridge, California
  - Alameda County Medical Center, Oakland, California
  - Health Management Institute, Inc., San Francisco, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente, Denver, Colorado
  - Blick Medical Associates, Norwalk, Connecticut
  - Biogenomx Research Institute, LLC, Fort Lauderdale, Florida
  - Life Way Inc., Fort Lauderdale, Florida
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - HIV Clinical Research, Fort Lauderdale, Florida
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - University of Florida, Jacksonville, Florida
  - The Kinder Medical Group, Miami, Florida
  - University of Miami, Miami, Florida
  - South Florida Infectious Diseases and Tropical Medicine Center, Miami, Florida
  - Community Health of South Florida Inc., Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Diseases Associates of NW FL, Pensacola, Florida
  - Associates in Infectious Diseases, Port Saint Lucie, Florida
  - Barry M. Rodwick, M.D., Safety Harbor, Florida
  - USF Health, Tampa, Florida
  - Infectious Disease Research Institute, Inc., Tampa, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - Atlanta Infectious Disease Group, PC, Atlanta, Georgia
  - Infectious Disease Solutions, Atlanta, Georgia
  - Family Healthcare of Atlanta PC, Atlanta, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - NorthStar Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Chase Brexton Health Services, Baltimore, Maryland
  - MetroWest Medical Center, Framingham, Massachusetts
  - Community Research Initiative of New England - WEST, Springfield, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, College of Osteopathic Medicine, East Lansing, Michigan
  - St. John Hospital Internal Medicine Clinic - Mack Office Building, Grosse Point Woods, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - ID Associates, PA, Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Upstate Infectious Diseases Associates, Albany, New York
  - Greiger Clinic, Mount Vernon, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - AIDS Community Health Center, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - ID Consultants, P.A., Charlotte, North Carolina
  - East Carolina University The Brody School of Medicine, Greenville, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Summa Health System Care Center, Akron, Ohio
  - Central Texas Clinical Research, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - North Texas Inf. Disease Consultants, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Valley AIDS Counsel, Harlingen, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon E. Crofoot, MD, PA, Houston, Texas
  - Daniel Coulston, MD, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - Canadian Immunodeficiency Research Collaborative Incorporated, Toronto, Ontario
  - CascAids Research, Toronto, Ontario
  - Clinique Du Quartier Latin, Montreal, Quebec
- Puerto Rico (3):
  - Instituto de Investigacion Cientifica del Sur, Ponce
  - Clinical Research Puerto Rico Inc, San Juan
  - University of Puerto Rico, San Juan

REFERENCES:
- [Derived] Campo R, DeJesus E, Bredeek UF, Henry K, Khanlou H, Logue K, Brinson C, Benson P, Dau L, Wang H, White K, Flaherty J, Fralich T, Guyer B, Piontkowsky D. SWIFT: prospective 48-week study to evaluate efficacy and safety of switching to emtricitabine/tenofovir from lamivudine/abacavir in virologically suppressed HIV-1 infected patients on a boosted protease inhibitor containing antiretroviral regimen. Clin Infect Dis. 2013 Jun;56(11):1637-45. doi: 10.1093/cid/cis1203. Epub 2013 Jan 29. PMID 23362296
- See also: Click here for more information about Truvada — http://www.truvada.com
- See also: Gilead Website — http://www.gilead.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 76 study sites; 70 in the US, 3 in Canada, and 3 in Puerto Rico. The first participant was screened on 15 August 2008, and the last participant was randomized on 27 April 2010. Last participant observation (LPO) date was 19 April 2011
Pre-assignment Details: A total of 393 subjects were screened for entry into this study, and 312 subjects were randomized (156 to each treatment group). One participant randomized to the TVD+PI/r group was never treated.
Groups:
- FTC/TDF (Truvada [TVD]) + PI/r (Ritonavir-boosted PI Regimen): Participants in this group received fixed-dose combination FTC 200 mg/TDF 300 mg (Truvada [TVD]) for 48 weeks. The participant's prestudy ritonavir-boosted PI was continued unmodified through the 48 weeks of the study.
- Abacavir (ABC) /Lamivudine (3TC) + PI/r (Ritonavir-boosted PI): Participants in this group continued their prestudy therapy - ABC 600 mg/3TC 300 mg administered as one tablet orally once daily (Epzicom) plus ritonavir-boosted PI regimen, given orally for 48 weeks.
Period: Overall Study
Arm/Group | FTC/TDF (Truvada [TVD]) + PI/r (Ritonavir-boosted PI Regimen) | Abacavir (ABC) /Lamivudine (3TC) + PI/r (Ritonavir-boosted PI)
Started | 155 | 156
Completed | 138 | 139
Not Completed | 17 | 17
Not completed — Adverse Event | 7 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Lost to Follow-up | 4 | 5
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TVD + PI/r: Participants in this group received fixed-dose combination FTC 200 mg/TDF 300 mg (Truvada [TVD]) for 48 weeks. The participant's prestudy ritonavir-boosted PI was continued unmodified through the 48 weeks of the study.
- Total: Total of all reporting groups
Arm/Group | TVD + PI/r | ABC/3TC + PI/r | Total
Number analyzed (Participants) | 155 | 156 | 311
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (9.0) | 47 (9.7) | 46 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 129 | 134 | 263
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 44 | 87
  White | 96 | 106 | 202
  Other | 12 | 3 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 38 | 36 | 74
  Non-Hispanic/Latino | 117 | 120 | 237
Region of Enrollment [Number; unit: participants]
  United States | 146 | 142 | 288
  Puerto Rico | 4 | 5 | 9
  Canada | 5 | 9 | 14
Weight [Mean (Standard Deviation); unit: kg] | 82.2 (17.40) | 82.5 (15.65) | 82.3 (16.52)
Height [Mean (Standard Deviation); unit: cm] | 173.8 (9.52) | 174.1 (9.55) | 173.9 (9.52)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (5.96) | 27.2 (4.93) | 27.3 (5.46)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 Ribonucleic Acid (RNA) < 200 Copies/mL Through Week 48 Based on Time to Loss of Virologic Response (TLOVR) Algorithm
Description: The percentage of participants with HIV-1 RNA < 200 copies/mL based on TLOVR algorithm at Week 48 was summarized. Participants were considered nonresponders in the TLOVR analysis if they experienced virologic rebound prior to or at Week 48, discontinued study before Week 48, or added a new antiretroviral (ARV) agent prior to completion of the study. Virologic rebound was defined as 2 consecutive HIV-1 RNA values >= 200 copies/mL or the last HIV-1 RNA value >= 200 copies/mL followed by discontinuation from the study.
Time Frame: Baseline to 48 weeks
Population: Intent-to-treat (ITT) Analysis Set: Participants who were treated with at least one dose of study drug with no documented resistance to study drug prior to screening.
Measure: Number; unit: percentage of participants
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 154 | 156
percentage of participants | 86.4 | 83.3
Statistical Analysis 1: Comparison: TVD + PI/r vs ABC/3TC + PI/r; Null hypothesis: The TVD group is at least 12% worse than the ABC/3TC group with respect to the percentage of subjects maintaining HIV-1 RNA < 200 copies/mL through Week 48 ("responder rate", as defined by the TLOVR algorithm) Alternative hypothesis: The TVD group is less than 12% worse than the ABC/3TC group with respect to the percentage of subjects maintaining HIV-1 RNA < 200 copies/mL through Week 48 ("responder rate", as defined by the TLOVR algorithm); Test type: Non-Inferiority or Equivalence — This study was designed to show noninferiority (change of < 12%) in regard of proportions of responders (TLOVR) at Week 48. With 170 subjects in each group, the lower limit of observed one-sided 97.5% confidence interval was expected to be greater than -0.120 with 80% power when the proportion of responders in both treatment groups is 0.820 (82%) at Week 48. 312 subjects were enrolled, representing 8% less than planned (n = 340). As a result, power to claim non-inferiority decreased to 78%; Inverted two one-sided tests; Inverted two one-sided tests with the standardized statistic; Difference in percentages between groups = 3.0, 95% CI 2-sided [-5.1 to 11.2]

2. Secondary Outcome: Percentage of Participants With Pure Virologic Response (PVR) for HIV-1 RNA Cutoff at 200 Copies/mL Through Week 48
Description: The percentage of participants with PVR for HIV-1 RNA cutoff at 200 copies/mL at Week 48 was summarized. Pure virologic response was the percentage of subjects who did not have a virologic rebound. Virologic rebound was defined as two consecutive HIV-1 RNA values >= 200 copies/mL or the last HIV-1 RNA value >= 200 copies/mL followed by discontinuation from the study.
Time Frame: Baseline to 48 weeks
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 154 | 156
percentage of participants | 99.2 [94.8 to 99.9] | 97.2 [92.7 to 98.9]

3. Secondary Outcome: Percentage of Participants With Pure Virologic Response (PVR) for HIV-1 RNA Cutoff at 50 Copies/mL Through Week 48
Description: The percentage of participants with PVR for HIV-1 RNA cutoff at 50 copies/mL at Week 48 was summarized. Pure virologic response was the proportion of participants who did not have a virologic rebound. Virologic rebound was defined as two consecutive HIV-1 RNA values >= 50 copies/mL or the last HIV-1 RNA value >= 50 copies/mL followed by discontinuation from the study.
Time Frame: Baseline to 48 weeks
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 154 | 156
percentage of participants | 93.0 [87.3 to 96.2] | 91.1 [85.1 to 94.7]

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 200 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA < 200 copies/mL at Week 48 was summarized.
Time Frame: 48 weeks
Population: ITT analysis set
  Missing = Failure: Participants with missing values considered to have HIV-1 RNA levels >= 200 copies/mL
  Virologic Success: Last available HIV-1 RNA < 200 copies/mL in the Week 48 window while on randomized treatment
Measure: Number; unit: percentage of participants
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 154 | 156
percentage of participants
  On-Treatment Response Analysis (Missing = Failure) | 84.4 | 82.1
  Snapshot Responder Analysis (Virologic Success) | 84.4 | 82.1

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was summarized.
Time Frame: 48 weeks
Population: ITT analysis set
  TLOVR: No virologic rebound on or before Week 48; no discontinuation before Week 48; no new ARV by study completion
  Missing = Failure: Participants with missing values considered to have HIV-1 RNA levels >= 50 copies/mL
  Virologic Success: Last available HIV-1 RNA < 50 copies/mL in Week 48 window on randomized treatment
Measure: Number; unit: percentage of participants
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 154 | 156
percentage of participants
  TLOVR Responder Analysis | 77.9 | 76.3
  On-Treatment Response Analysis (Missing = Failure) | 79.9 | 77.6
  Snapshot Responder Analysis (Virologic Success) | 79.9 | 77.6

6. Secondary Outcome: Change From Baseline in Cluster Determinant 4 (CD4) Cell Count at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: ITT Analysis Set
  Missing = Excluded: Participants with missing values were excluded from this analysis
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 135 | 138
cells/microliter | 8 (148.3) | 34 (150.1)

7. Secondary Outcome: Change From Baseline Calculated Creatinine Clearance (CLcr) Using Ideal Body Weight by Cockcroft-Gault Method at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set: The treated analysis set included all randomized participants who received at least one dose of study drug. Participants who were randomized to continue ABC/3TC+PI/r during the study were included in the treated analysis set if they took at least one dose of their study drug after the baseline visit.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 137 | 139
mL/min | -8.4 (12.18) | -4.1 (12.99)

8. Secondary Outcome: Change From Baseline Estimated Glomerular Filtration Rate (eGFR) by Modified Diet in Renal Disease (MDRD) at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 137 | 139
mL/min/1.73m^2 | -9.0 (14.10) | -3.7 (15.75)

9. Secondary Outcome: Change From Baseline Fasting Glucose at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 134 | 135
mg/dL | 1 (23.1) | 1 (16.8)

10. Secondary Outcome: Change From Baseline Fasting Lipid Parameters at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 135 | 136
mg/dL
  Total Cholesterol | -21 (38.6) | -4 (37.9)
  LDL (low-density lipoprotein) | -6 (33.2) | 2 (30.0)
  HDL (high-density lipoprotein) | -2 (10.7) | 0 (11.3)
  Triglycerides | -51 (174.0) | -23 (178.3)

11. Secondary Outcome: Change From Baseline Ratio of Fasting Total Cholesterol Over High-density Lipoprotein (HDL) Cholesterol at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 135 | 136
Ratio | -0.1 (2.58) | -0.1 (1.03)

12. Secondary Outcome: Change From Baseline C-Reactive Protein at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set, Subset of Subjects Enrolled after Amendment 3
  Missing = Excluded
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 69 | 57
mg/dL | -0.026 (0.4029) | 0.225 (1.2787)

13. Secondary Outcome: Change From Baseline Fibrinogen at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set, Subset of Subjects Enrolled after Amendment 3
  Missing = Excluded
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 64 | 56
mg/dL | -4 (77.0) | 14 (91.8)

14. Secondary Outcome: Change From Baseline Interleukin-6 (IL-6), Interleukin-10 (IL-10), and Tumor Necrosis Factor-alpha (TNF-alpha) at Week 48
Description: Change = Week 48 value minus baseline value
Time Frame: Baseline to 48 weeks
Population: Treated Analysis Set, Subset of Participants Enrolled after Amendment 3
  Missing = Excluded
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Number analyzed (Participants) | 68 | 56
pg/mL
  IL-10 | 0.0 (1.69) | -0.2 (1.41)
  IL-6 | -0.2 (4.10) | -0.6 (5.96)
  TNF-alpha | 0.0 (2.06) | 4.7 (23.95)

ADVERSE EVENTS:
Time Frame: AEs were reported in the during the randomized, open-label study period between Weeks 0 through 48.
Arm/Group | TVD + PI/r | ABC/3TC + PI/r
Serious Adverse Events (participants affected / at risk) | 12/155 | 11/156
Other Adverse Events (participants affected / at risk) | 35/155 | 32/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TVD + PI/r (N=155) | ABC/3TC + PI/r (N=156)
Myocardial Infarction (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 0
Giardiasis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Streptococcal Sepsis (Infections and infestations) | 1 | 0
Shunt Infection (Infections and infestations) | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 0
Burns Third Degree (Injury, poisoning and procedural complications) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Hallucination, Auditory (Psychiatric disorders) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TVD + PI/r (N=155) | ABC/3TC + PI/r (N=156)
Diarrhea (Gastrointestinal disorders) | 13 | 11
Upper Respiratory Tract Infection (Infections and infestations) | 14 | 14
Headache (Nervous system disorders) | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years